CLINICAL TRIAL: NCT03812835
Title: A PHASE IV NON-INTERVENTIONAL STUDY. REGISTRY OF ADVERSE EVENTS (AES)/SUSPECTED ADVERSE DRUG REACTIONS (SADRS) OF ADULT PATIENTS UNDER TREATMENT OF DEEP VEIN THROMBOSIS (DVT) AND PULMONARY EMBOLISM (PE); PREVENTION OF RECURRENT DVT AND PE WITH ELICUIS REGISTERED (APIXABAN)
Brief Title: A Study of Adverse Events and Suspected Adverse Drug Reactions of Patients Under Treatment of Apixaban for Venous Thomboembolism (VTE) Treatment
Status: Withdrawn | Type: Observational
Why Stopped: Company decision to not conduct study and was cancelled prior to any enrollment.
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: B0661104
Record Dates: First submitted 2019-01-04; First posted 2019-01-23 (Actual); Last update posted 2021-11-11 (Actual); Status verified 2021-11

CONDITIONS: Thrombosis, Deep Vein; Pulmonary Embolism
MeSH Terms: conditions — Venous Thrombosis; Pulmonary Embolism

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective

SUMMARY:
Number, type and incidence of adverse events/suspected adverse drug reactions in patients treated with apixaban, according to therapeutic indications approved in Mexico.

ELIGIBILITY:
Inclusion Criteria:

Patients must meet all of the following inclusion criteria to be eligible for inclusion in the study:

1. Evidence a personally signed and dated informed consent document indicating that the patient (or a legally acceptable representative) has been informed of all pertinent aspects of the study.
2. Patients (men and women) >18 years old.
3. Patients who have received at least one dose of apixaban for treatment of deep vein thrombosis (DVT) and pulmonary embolism (PE); prevention of recurrent DVT and PE

   -

Exclusion Criteria:

Patients meeting any of the following criteria will not be included in the study:

1. Patients who are participating in a clinical trial.
2. Hypersensitivity to the active substance or to any of the excipients.
3. Active clinically significant bleeding.
4. Hepatic disease associated with coagulopathy and clinically relevant bleeding risk, based on hepatic function tests.
5. Lesion or condition if considered a significant risk factor for major bleeding. This may include current or recent gastrointestinal ulceration, presence of malignant neoplasms at high risk of bleeding, recent brain or spinal injury, recent brain, spinal or ophthalmic surgery, recent intracranial hemorrhage, known or suspected esophageal varices, arteriovenous malformations, vascular aneurysms or major intraspinal or intracerebral vascular abnormalities.
6. Concomitant treatment with any other anticoagulant agent e.g. unfractionated heparin (UFH), low molecular weight heparins (enoxaparin, dalteparin, etc.), heparin derivatives (fondaparinux, etc.), and oral anticoagulants (warfarin, acenocoumarin, rivaroxaban, dabigatran, etc.) except under specific circumstances of switching anticoagulant therapy.
7. Pregnancy and breast-feeding.
8. Severe acute or chronic psychiatric condition and other significant medical condition.

   -

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients who have received at least one dose of apixaban for treatment of deep vein thrombosis (DVT) and pulmonary embolism (PE); prevention of recurrent DVT and PE.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2021-08-23 (Estimated); Primary Completion 2023-08-23 (Estimated); Study Completion 2023-08-23 (Estimated)

PRIMARY OUTCOMES:
The number, type and incidence of adverse events/suspected adverse drug reactions in patients treated with apixaban, according to therapeutic indications approved in Mexico. | 12 up to 24 months
  Data will be collected for at least 12 months and until 24 months in 3 sites in Mexico using an electronic case report form

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.